CLINICAL TRIAL: NCT06255431
Title: EFFECTIVENESS AND SAFETY OF CREAM CONTAINING SPENT GRAIN WAX EXTRACT, ARGAN OIL, AND SHEA BUTTER POST-TRICHOLOROACETIC ACID 15% PEEL: RANDOMIZED, CONTROLLED, DOUBLE-BLIND, SPLIT-FACE CLINICAL TRIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dina Kusumawardhani, dr., Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-02-0295
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Aging Disorder
Keywords: aging; skin aging; trichloroacetic acid; chemical peel; anti-inflammation; moisturizer

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, double-blinded, split face trial on women undergoing TCA 15% chemical peels.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cream Containing Spent Grain Wax Extract, Argan Oil, and Shea Butter (Ezerra Cream) (Active Comparator): Ezerra cream The creams are applied to the face twice daily (0,5 Finger Tip Unit/FTU), immediately after washing.
  group A (intervention cream on the right side of the face and control cream on the left side of the face) and group B (intervention cream on the left side of the face and control cream on the right side of the face).
  Interventions: Drug: Ezerra cream
- Vehicle cream (Placebo Comparator): Vehicle cream was prepared by the Pharmacy Department of Faculty of Medicine Universitas Indonesia and has similar consistency, color, and scent as the intervention cream. The creams are applied to the face twice daily (0,5 Finger Tip Unit/FTU), immediately after washing.
  Interventions: Drug: Ezerra cream

INTERVENTIONS:
Drug: Ezerra cream — The research subjects were divided into 2 groups: group A (intervention cream on the right side of the face and control cream on the left side of the face) and group B (intervention cream on the left side of the face and control cream on the right side of the face).
  The test material consists of a cream containing a mixture of spent grain wax extract, shea butter, and argan oil, along with a vehicle cream. Vehicle cream was prepared by the Pharmacy Department of Faculty of Medicine Universitas Indonesia and has similar consistency, color, and scent as the intervention cream.The creams are applied to the face twice daily (0,5 FTU), immediately after washing, in equal amounts on each side of the face. The creams are applied for 7 days, and participants are instructed to use appropriate sunscreen.
  Other Names: Vehicle cream

SUMMARY:
Chemical peels are resurfacing procedures where chemical agent causes controlled exfoliation of the skin, followed by regeneration and remodelling of the epidermis and dermis layers. Chemical peels can be used to treat various skin condition, such as skin aging, pigmentary disorders, and skin texture disorders. The use of moisturizer after chemical surgery can help speed up the wound healing process and repair the skin barrier. TCA chemical peel has more side effects than other chemical peel solutions. The risk of complications after TCA chemical surgery on Fitzpatrick IV-VI skin types is also higher, especially post-inflammatory hyperpigmentation. There is no specific recommendations regarding the type of moisturizer that can be used after TCA chemical peels. This study aims to assess the effectiveness of a cream containing spent grain wax, argan oil, and shea butter in reducing TCA peel side effects.

ELIGIBILITY:
Inclusion Criteria:

women, 30 - 60 years old with facial skin aging underwent chemical peeling with TCA 15%, have received priming with topical retinoic acid 0.05%, for at least 2 weeks and its use has been discontinued three days before chemical peel.

Exclusion Criteria:

Pregnant or lactating women, patients who received hormonal therapy, immunosuppressants, allergic to any of treatment ingredients, had active skin diseases on the face (acne vulgaris, seborrheic dermatitis, dll), history of keloid/hypertrophic scar, open wound, active infection, or history of recurrent herpes simplex

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 27 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss | Baseline (30 minutes after peeling), day 3, and day 7
Skin Capacitance | Baseline (30 minutes after peeling), day 3, and day 7
Erythema index | Baseline (30 minutes after peeling), day 3, and day 7

SECONDARY OUTCOMES:
global investigator assessment | Baseline (30 minutes after peeling), day 3, and day 7
  comprised individual ratings of erythema, desquamation, edema, each on 4-point-scale (0-None; 1-Mild; 2-Moderate, 3-Severe
subject self-assessment | Baseline (30 minutes after peeling), day 3, and day 7
  comprised individual ratings of erythema, desquamation, burning, pain, and itch, each on a 4-point-scale (0-None; 1-Mild; 2-Moderate, 3-Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kusumawardhani, Principal Investigator — Indonesia University
Locations (1):
- Faculty of Medicine Universitas Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided